CLINICAL TRIAL: NCT04832477
Title: PrEP Connected Study
Brief Title: Assessing the PrEP Care Cascade Among Black Men and Transwomen in the Southeastern US
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Lisa Eaton, Professor, University of Connecticut
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H20-0117
Record Dates: First submitted 2021-03-29; First posted 2021-04-05 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: HIV Seropositivity; Substance Use; STI; Stigma, Social
MeSH Terms: conditions — HIV Seropositivity; Substance-Related Disorders; Sexually Transmitted Diseases; Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stigma Counseling for PrEP Access (Other): Behavioral counseling
  Interventions: Behavioral: Stigma counseling for PrEP use

INTERVENTIONS:
Behavioral: Stigma counseling for PrEP use — This counseling consists of a single-session (45 minute) delivered by trained peer counselors. The primary aims and relevant content areas for counseling are: (1) Assessing and discussing factors known to be drivers of emotional barriers to accessing health care. This counseling aim has two main sub-components: (a) participants will be asked about their prior experiences with accessing health care and their concerns regarding future access, and (b) the counseling will focus on creating personal agency around needing to prioritize one's health. (2) Evaluating concerns around discussing PrEP with health care providers. The counseling combines motivational interviewing with medical decisional balance, which focuses on points to consider when evaluating PrEP. (3) Promoting resiliency beliefs and positive adaptation. For this objective the counselor works with the participant to establish PrEP use goals and problem-solving strategies.

SUMMARY:
The proposed research aims to assess the multiple forms and paths of stigma and substance use as they relate to pre-exposure prophylaxis (PrEP) use for HIV prevention. How stigma and an evolving public health landscape impact PrEP use among Black sexual minorit men who use substances is unknown. The current application focuses on addressing critical and novel questions to improving the essential building blocks of biomedical prevention approaches by providing crucial information for enhancing interventions to lower HIV prevalence among substance using Black sexual minority men.

DETAILED DESCRIPTION:
HIV incidence among Black men who have sex with men (BMSM) in the southeastern United States is one of the highest in the world. Our research team has conducted studies with BMSM in Atlanta that have demonstrated 35% HIV prevalence and over 5% annual HIV incidence. Although PrEP is highly effective for preventing HIV transmission, it is not reaching BMSM. The failures in our ability to engage BMSM in PrEP use are highly problematic given the alarming rates of HIV transmission among this group. Of particular concern is the impact of substance use as a barrier in PrEP linkage, uptake, adherence, and persistence. Substance use is common among BMSM in our study, with 43% (n=204/474) reporting recent substance use. Further complicating PrEP use is the potential impact of COVID-19 on health care access, health care infrastructure, and sex behavior. The need to better understand PrEP use in the context of our new health care landscape is critical to making advances in PrEP use. At this point, assessing how substance use impacts PrEP use is challenging because PrEP implementation is so low among this group. The current study aims to provide substance using BMSM with evidence-based PrEP engagement counseling to address barriers to accessing PrEP (not for intervention testing, but for facilitating PrEP use) and to assess the multiple forms and paths of stigma and substance use as they relate to PrEP linkage, uptake, adherence, and persistence. The investigators propose using the HIV Stigma Framework as a conceptual model for investigating the intersecting pathways of stigma drivers and stigma mechanisms as they relate to PrEP use among substance using BMSM. Aim 1: Enroll a prospective cohort of N=500 BMSM who test HIV negative and test substance use positive on toxicology testing, and provide evidence-based PrEP engagement counseling to facilitate access to PrEP care. Aim 2: Conduct psychosocial and health care access assessments every 2-months for 18-months, and conduct HIV/STI testing and dried blood spot testing for TFV-DP every 3-months for 18-months. Aim 3: Using data collected from Aims 1 and 2, model stigma pathways of advancing and reverting along the PrEP cascade (i.e., linkage, uptake, adherence, persistence), with these pathways mediated by health care access and moderated by substance use. Achieving the aims will provide critical insight for translating and adapting interventions to enhance potency and durability for individuals at exceedingly elevated risk for HIV.

ELIGIBILITY:
Inclusion Criteria:

* Men (based on male sex assignment at birth)
* Age 18 or older
* Identify as Black, African-American, Afro-Brazilian, Afro-Carribean, or African diaspora,
* Report condomless anal sex with man in past six months
* Test HIV negative
* Report recent (<3 months) substance use
* Positive drug toxicology for substance use

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2026-02-04 (Estimated); Study Completion 2026-02-04 (Estimated)

PRIMARY OUTCOMES:
PrEP Use | 12 months
  TFV-DP (Tenofovir Diphosphate) biological testing for PrEP pill taking will be assessed. TFV-DP measured at >700 fmol will be interpreted as having taken ≥4 doses/week, and TFV-DP measured at >700 fmol over two consecutive time points will be interpreted as persistence to taking PrEP. The lower scale limit is 0 and upper scale limit is approximately around 2500. Higher values indicate greater medication adherence to PrEP pills.

SECONDARY OUTCOMES:
PrEP stigma | 12 months
  Questionnaire to assess stigma related psychosocial variables will be used to assess secondary outcomes. This questionnaire is based measures provided in the HIV Stigma Framework for assessing HIV related stigma (i.e., prejudice, stereotypes, discrimination, enacted stigma, anticipated stigma, and internalized stigma). Responses to the scale items range from 1=strongly disagree to 6=strongly agree, with higher scores indicating a higher number of experiences of stigma.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Eaton, PhD, Principal Investigator — University of Connecticut
Locations (1):
- SHARE Project, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No